#### RESEARCH INFORMATION SHEET

Dear. Mr / Mrs / Brothers / Sisters

With this we explain that Tuberculosis (TB) is a disease that attacks various organs, especially the lungs. One of the complications of TB disease is Tuberculosis Meningitis, this disease can reduce the quality of life of the sufferer, such as malnutrition (malnutrition and vitamin D deficiency). For that we will conduct a study for four weeks (28 days) on Mr / Mrs / Brother / i to be able to improve the condition of Mr / Mrs / Brother / i by providing porridge high in protein, calcium and vitamin D. If Mr / Mrs / Brother / i are willing to take part in this research, then:

- 1. Interview about: age and gender
- 2. Interview about food and beverages by interviewing eating habits once, namely at the beginning of the week.
- 3. Blood draw  $\pm$  3 mL or one teaspoon which is done 2 times, namely at the beginning of the week and the end of the week to determine the level of vitamin D and several tests that affect the condition of the disease

As a result of taking blood, you may feel some discomfort or pain, but this can be minimized by taking blood by trained personnel and using a small syringe.

The participation of Mr / Mrs / Brothers / Sisters in this research is voluntary and Mr / Mrs / Brother / i can refuse or resign during the research process.

The advantage for Mr / Mrs / Brothers / Sisters if you participate in this research is that you can find out the state of health and nutrition and know the levels of vitamin D. All data in this study are confidential.

If Mr / Mrs / Brothers / Sisters are willing to participate in this research, then we will ask for his willingness to be able to sign a letter of approval to become research participants:

# UTILIZATION OF HIGH INTAKE OF PROTEIN, VITAMIN D, AND CALCIUM AS MARKERS OF BIOMOLECULAR IMPROVEMENT IN TUBERCULOSIS AND COMPLICATIONS

Things that are not clear in this study can be asked directly or by telephone to the person in charge of this research, namely Prof. Dr. dr. Dina Keumala Sari, MG. SpGK through the Department of Nutrition, FK USU, house: ring road, komp. Tasbih 2, block 5. Number 126, Medan, North Sumatra, Indonesia, telephone: 061-4256-4286, cell phone: 081397177693. For the willingness of Mr / Mrs / Brothers / Sisters, thank you.

### **Informed Consent**

### FACULTY OF MEDICINE UNIVERSITAS SUMATERA UTARA

## LETTER OF AGREEMENT TO BE A RESEARCH PARTICIPANT

I, the undersigned below:

| Name | : | | |
|---|---|---|---|
| Age | : | | |
| Gender | : Male / Female | | |
| Address | : | | |
| After receiving suffic | eient information and underst | anding the benefits | of the research below, |
| entitled: | | | |
| | TION OF HIGH INTAKE (<br>AS MARKERS OF BIOMO)<br>TUBERCULOSIS AND C | LECULAR IMPR | OVEMENT IN |
| Voluntarily agreeing to be included in the above research provided that at any time you are | | | |
| harmed in any form h | as the right to cancel this agre | ement. | |
| Mengetahui: | | Medan, | 2019 |
| Who responsible for research: | | Who approved | |
| (Prof. Dr. dr. Dina Ke | eumala Sari, MG. Sp. GK ) | ( | ) |
| The Witness | 3: | | |
| ( | ) | | |